CLINICAL TRIAL: NCT01896076
Title: The Caudal Space in Children: Ultrasound Evaluation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0244
Record Dates: First submitted 2013-06-30; First posted 2013-07-11 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Hydrocele; Inguinal Hernia; Hypospadia; Cryptorchidism; Genitourinary Disease
Keywords: caudal space; children; ultrasound evaluation
MeSH Terms: conditions — Testicular Hydrocele; Hernia, Inguinal; Hypospadias; Cryptorchidism; Urogenital Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric patients in urologic surgery: Pediatric patients undergoing caudal block for urologic surgery were included in this study.
  Interventions: Other: ultrasound evaluation of caudal space

INTERVENTIONS:
Other: ultrasound evaluation of caudal space — After induction of general anesthesia, the patients were placed in the lateral position. The ultrasound evaluation include transverse and longitudinal view.
  First, investigators place the transducer at the sacral cornua to obtain a transverse view.
  In the transverse view, the distance between two cornua and the depth of caudal space at the sacral hiatus were measured. In the longitudinal view, the distance from the skin to the sacrococcygeal membrane and the optimal angles and the safety distance for needle insertion depending on the points of insertions were measured. From the end of dura sac to the sacral hiatus were regarded as safety distance for the needle insertion during caudal block.

SUMMARY:
Caudal anesthesia is commonly employed in pediatrics to produce postoperative analgesia in low abdominal or urologic surgery.

An exact understanding of the anatomy of the sacral area including sacral hiatus and surrounding structures is crucial to the success of caudal block.

The aim of this study is to evaluate the anatomy of the caudal space in pediatrics by ultrasound evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 - 84 months who were scheduled to undergo elective urological surgery.

Exclusion Criteria:

* Patients with any contraindication to caudal epidural block were excluded.

  * coagulopathy
  * allergy to local anesthetics
  * infection at the puncture site

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 0 - 84 months who were scheduled to undergo elective urological surgery. This investigation was conducted at a single tertiary medical center (Severance Hospital), Seoul, Republic of Korea.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
ultrasound evaluation of caudal space | Right after induction of general anesthesia, the patients were placed in the lateral position. The ultrasound evaluation include transverse and longitudinal view.
  First, investigators place the transducer at the sacral cornua to obtain a transverse view.
  In the transverse view, the distance between two cornua and the depth of caudal space at the sacral hiatus were measured. In the longitudinal view, the distance from the skin to the sacrococcygeal membrane and the optimal angles and the safety distance for needle insertion depending on the points of insertions were measured. From the end of dura sac to the sacral hiatus were regarded as safety distance for the needle insertion during caudal block.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea